CLINICAL TRIAL: NCT05969327
Title: Role of Vitamin D Therapy in Recovery From Early Neonatal Sepsis (Randomized Controlled Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MD 438/ 2017
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2017-12

CONDITIONS: Importance of Vitamin D Therapy in Treatment of Neonatal Sepsis
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- with out vitamin D (No Intervention): neonates without supplementation
- Vitamin D 400 IU (Experimental): neonates with 400 IU supplementation
  Interventions: Drug: Vitamin D
- Vitamin D 800 IU (Experimental): neonates with 800 IU supplementation
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — oral supplementation of two different doses
  Arms: Vitamin D 400 IU; Vitamin D 800 IU

SUMMARY:
Neonatal sepsis is still a major cause of morbidity and mortality despite major advances in neonatal intensive care units. Early-onset sepsis (EOS) is an infection of the blood acquired vertically from the mother and manifests shortly after birth. The objective of this study is to assess the vitamin D status in neonates with Early onset sepsis (EOS) and evaluate the influence of different doses of vitamin D3 (800 IU/d versus 400 IU/d), in these infants.

DETAILED DESCRIPTION:
Subjects:

This is a randomized controlled trial (RCT) conducted on sixty (66) full term newborns with clinical and laboratory findings of early onset of sepsis (EOS) and admitted to the Neonatal Intensive Care Unit of El-Demerdash hospital of Ain Shams university and El Ahrar teaching hospital in Zagazig.

* Inclusion Criteria: full term newborns with clinical and laboratory findings of early onset of sepsis (EOS).
* Exclusion Criteria: Preterm newborn, NPO neonates , infants with maternal risk factors , such as clinical and/or histological chorioamnionitis, neonates delivered at home ,neonates to mothers with premature rupture of membrane, and major congenital abnormalities which may be predisposing factors for development of EOS.

NB: we excluded the dead cases (6 cases) in the final laboratory and clinical relation with serum Vitamin D levels after recovery because sepsis caused death to these neonates and recovery didn't occur .

Methods:

An informed consent was taken from the legal guardian of the newborns participating in the study.

Detailed history taking from all mothers of neonates in the study laying stress on vitamin D supplementation during pregnancy, sun exposure in mothers during pregnancy, place and mode of delivery. Dietetic history in all included mothers (National Nutrition institute, 2006). Clinical evaluation of all newborns for signs of neonatal sepsis.

All subjects in the study were subjected to the following:

1. Clinical Examination: General examination including vital data; temperature, pulse, respiratory rate, anthropometric measurements including weight and length (Neonatal Anthropometry): In all neonates weight (in Kg) was recorded on an electronic weighing scale at birth. Length (in cm) was recorded by measuring tape.

   SDS of weight and length was calculated and plotted against appropriate growth curves (Tanner et al., 1968).
2. Laboratory Investigations: Under aseptic conditions venous blood samples was collected into sterile blood collection tubes and the following investigations was performed:

   * A neonatal sepsis screen including: total leukocyte count, absolute neutrophil count, platelet count immature to total neutrophil count and C-reactive protein (CRP).
   * Blood samples for complete blood count (CBC) and blood culture. All patients were initially assessed according to Newborn Scale of Sepsis.

     * A total clinical score less than 10 indicated that the newborn did not have sepsis-a negative predictive value of 97%.
     * Any neonate with a total clinical score greater than 10 was considered ''sick,'' possibly with sepsis. A clinical score greater than 10 is also an indicator of the need for further diagnostic evaluation (Gardner, 2008).
   * Serum 25 (OH) vitamin D levels: was measured by Human Vitamin D ELISA Kit (Qualpro diagnostics, INDIA) in all newborns on the first day of sepsis, 25(OH) vitamin D levels were classified according to the guidelines of the Endocrine Society to the following reference values:
   * Sufficient >20 ng/ml (>50 nmol/l)
   * Insufficient 12-20 ng/ml (30-50 nmol/l)
   * Deficient <12 ng/ml (<30 nmol/l) (Munns et al., 2016).

Study design : Subjects were classified into three groups :

GROUP A (conventional dose Vitamin D) those neonates who received a daily dose of oral Vitamin D of 400 IU through Ryle or mouth from onset of diagnosis till recovery from sepsis.

GROUP B (higher dose Vitamin D) those neonates who receiveda daily dose of oral vitamin D of 800 IU through ryle or mouth from onset of diagnosis till recovery from sepsis.

GROUP C (Placebo group) those neonates with early onset sepsis who did not receive any vitamin D supplementation.

Patients were matched regarding sepsis score. All 3 groups were treated using strategy of sepsis treatment.

* Reevaluation of serum Vitamin D levels for all patients on recovery(recovery was assessed by Newborn Scale of Sepsis to be less than 10).
* Serum Ca and P were measured initially for all patients upon diagnosis of EOS, and on discharge upon recovery Normal range of Ca 8.8-11.3mg/dl Normal range P 4.5-6.2 mg/dl
* Urinary Ca will be evaluated after two weeks of onset of vitamin D therapy (for patients who experience elevation of serum Ca above normal value).

Type of Study: Randomized controlled study. Study Setting: This study was conducted on sixty (66) full term newborns with clinical and laboratory findings of early onset of sepsis (EOS) and were admitted to the Neonatal Intensive Care Unit of El-Demerdash hospital of Ain Shams university and El Ahrar teaching hospital in Zagazig.

* Study Period: The study took place from January 2018 to January 2021.
* Study Population: Full term newborns with early onset sepsis.
* Sampling Method: random.
* Sample Size:

Using PASS program, setting alpha error at 5% and power at 80%. After reviewing literature, no previous similar study has been done before. So assuming that NICU duration for placebo, 400IU vitamin D and 800 IU vitamin D respectively is 7±2.5, 5.5±2.5, 4±2.5 based on this, the needed sample is 20 cases per group (total 60).

• Ethical Considerations:

* The consent was conducted to the legal guardian or the parents of our patients by the investigator.
* Premature termination of oral vitamin D was mandatory for patients with abdominal distension or feeding intolerance.
* All data was treated confidentially and was not be allowed except to the principle investigator.

ELIGIBILITY:
Inclusion Criteria:

* -Inclusion Criteria: full term newborns with clinical and laboratory findings of early onset of sepsis (EOS).

Exclusion Criteria:

* Preterm newborn, NPO neonates , infants with maternal risk factors , such as clinical and/or histological chorioamnionitis, neonates delivered at home ,neonates to mothers with premature rupture of membrane, and major congenital abnormalities which may be predisposing factors for development of EOS.

Ages: 3 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Role of Vitamin D therapy in recovery from Early Neonatal Sepsis (randomized controlled trial) | nearly 4 years
  supplementation of Vitamin D

CONTACTS AND LOCATIONS:
Locations (1):
- Mayada Ahmad Mohamed, Zagazig, Egypt